CLINICAL TRIAL: NCT00005782
Title: Leukapheresis of Volunteers With Sickle Cell Trait to Evaluate Mobilization of Stem Cells With Granulocyte Colony-Stimulating Factor and Stem Cell Collection and Storage for Allogeneic Transplantation
Brief Title: Mobilization and Handling of Stem Cells for Transplant From Healthy Volunteers With Sickle Cell Trait
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000060; 00-DK-0060; NCT00001980 (obsolete NCT alias)
Record Dates: First submitted 2000-06-03; First posted 2000-06-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-07

CONDITIONS: Sickle Cell Trait
Keywords: Donor Apheresis; Sickle Cell Trait; Red Cell Alloimmunization
MeSH Terms: conditions — Sickle Cell Trait | interventions — Granulocyte Colony-Stimulating Factor; Leukapheresis

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor
Procedure: Leukapheresis

SUMMARY:
This study will examine the effects of granulocyte colony-stimulating factor (G-CSF) on bone marrow stem cells in healthy volunteers with sickle cell trait and determine if cells collected for transplantation from donors with sickle cell trait require special handling.

Stem cells, which the bone marrow produces, are responsible for making all the different kinds of blood cells. They are the cells used in bone marrow, or stem cell, transplantation. The drug G-CSF, which is a naturally occurring hormone, causes stem cells to mobilize-that is, to be released from the bone marrow and enter the blood stream. This drug is given to stem cell donors to increase the amount of cells that can be collected. Stem cell donors for patients with sickle cell disease are often healthy siblings of the patient who have a matching bone marrow type. Some siblings carry the sickle cell trait, however, and, even though they do not have sickle cell disease and their blood and bone marrow are normal, it is not known how their cells will react to G-CSF stimulation. Nor is it known if their stem cells require special methods of removal, processing or storing.

Healthy volunteers 18 years or older with sickle cell trait who have no history of sickle cell disease and no known medical problems may be eligible for this study. Participants will have a medical history and physical examination, including blood tests and urinalysis. They will receive injections of G-CSF under the skin once a day for 5 days. On the fifth day, stem cells will be collected through leukapheresis. In this procedure, whole blood is drawn from an arm vein, similar to donating whole blood. The blood then circulates through a cell separator machine, the stem cells are removed, and the rest of the blood is transfused back to the donor through a vein in the other arm.

The information gained from this study will be used to ensure the safety of stem cell donors with sickle cell trait and to better prepare stem cells for transplantation in sickle cell patients.

DETAILED DESCRIPTION:
Patients with sickle cell disease are increasingly becoming eligible for transplantation as the techniques of stem cell transplantation continue to improve, leading to less morbidity and mortality. However, the availability of a matched donor still remains one of the main obstacles. Given the inherited nature of this disease, many HLA-matched siblings of patients with sickle cell disease have sickle cell trait. Therefore, patients with sickle cell trait presumably have been used as donors for patients with sickle cell disease. However, there are no published data on whether special manipulations are required for the maintenance and storage of stem cells collected from patients with sickle cell trait. The effects of granulocyte-colony stimulating factor (G-CSF)-induced stem cell mobilization in these patients are also not known. Also, due to the potential of HbS gellation in red cells, the freezing of stem cells derived from individuals with sickle cell trait may require a more stringent red cell removal than is normally performed. We would like to evaluate these issues using volunteers with sickle cell trait prior to beginning our own transplant protocol for sickle cell disease.

ELIGIBILITY:
Confirmed diagnosis of sickle cell trait.

Greater than age 17.

No active systemic infection or history of recurrent infections requiring intravenous antibiotic treatment .

Normal renal function: creatinine less than 2X normal, or proteinuria less than 1+.

Normal liver function: bilirubin less than 2X normal, transaminases within normal limits.

Normal blood count: WBC 3,000-10,000/mm3, granulocytes greater than 1,500/mm3, platelets greater than 150,000/mm3, hemoglobin greater than 12.5g/dL, MCV and MCHC within normal limits.

Female volunteers of childbearing age should have a negative serum pregnancy test within one week of beginning G-CSF administration.

Eligible for normal blood donation (i.e. tested negative for syphilis (RPR), hepatitis B and C (Hasbro, Anti-Hubcap, Anti-HCV), HIV, and HTLV-1.

Subject must give informed consent to participate in the protocol.

No history of sickle cell crises.

Children less than 18 years of age are excluded as is per routine for normal volunteer protocols.

No active systemic viral, bacterial, fungal, or parasitic infection.

No female volunteers with positive pregnancy test or who are lactating.

No history of autoimmune disease, such as rheumatoid arthritis and systemic lupus erythematosus.

No history of cancer excluding squamous or basal cell carcinoma of the skin.

No history of any malignant hematologic disorders.

No history of cardiovascular disease or related symptoms such as chest pain and shortness of breath..

No allergy to G-CSF or bacterial E. coli products.

No history of G-CSF administration or leukapheresis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2000-01; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States